CLINICAL TRIAL: NCT03837873
Title: DLCL002 Protocol for Young Patients With Newly Diagnosed High Risk Aggressive B-cell Lymphoma, a Multicenter Phase II Study
Brief Title: DLCL002 Protocol for Patients With High Risk Aggressive B-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Principal Investigator, Zou Dehui, principal investigator, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2018010-EC-2
Record Dates: First submitted 2019-01-05; First posted 2019-02-12 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Diffuse Large B Cell Lymphoma; High-grade B-cell Lymphoma; Transformed Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Etoposide; Vincristine; Doxorubicin; Dexamethasone; Cyclophosphamide; Lenalidomide; Cisplatin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DLCL002 protocol (Experimental): Patients will receive R-DA-EDOCH(rituximab, etoposide, dexamethasone, vincristine, cyclophosphamide, doxorubicin) as induction therapy and be evaluated by PET CT after the fourth cycle. Patients achieve CR at interim-PET will receive either ASCT or the remaining 4 cycles of R-DA-EDOCH, while those achieve PR(Deauville score 4-5) will be rescued by two courses of R(2)-DHAP(rituximab, lenalidomide(only for patients with non-GCB DLBCL), dexamethasone, cisplatin, cytarabine). Patients who achieved CR+good PR(Deauville score 4) after the rescue therapy will be consolidated with ASCT,and those remain in PR(Deauville score 5) will receive other rescue treatments.
  Interventions: Drug: Rituximab; Drug: Etoposide; Drug: Vincristine; Drug: Doxorubicin; Drug: Dexamethasone; Drug: Cyclophosphamide; Drug: Lenalidomide; Drug: Cisplatin; Drug: Cytarabine

INTERVENTIONS:
Drug: Rituximab — rituximab 750mg/m2 i.v. on day 0
Drug: Etoposide — 50mg/m2, continuous i.v. on day 1-4
Drug: Vincristine — 0.4mg/m2, continuous i.v. on day 1-4
Drug: Doxorubicin — 10mg/m2, continuous i.v. on day 1-4
Drug: Dexamethasone — 30mg/day, i.v. on day 1-5 for R-DA-EDOCH regimen; 40mg/day, i.v. on day 1-4 for R(2)-DHAP regimen
Drug: Cyclophosphamide — 750mg/m2, i.v. on day5
Drug: Lenalidomide — 25mg/day, p.o. on day 0-9
Drug: Cisplatin — 100mg/m2 continuous i.v. on day 1
Drug: Cytarabine — 2g/m2 q12h, i.v. on day 2

SUMMARY:
Patients eligible for the study will receive R-DA-EDOCH as the induction therapy and be evaluated by PET CT after the fourth cycle. Patients achieve CR at interim-PET(Deauville score 1-3) will receive either ASCT or the remaining 4 cycles of R-DA-EDOCH, while those achieve PR(Deauville score 4-5) will be rescued by two courses of R(2)-DHAP and then be revaluated by the second interim-PET. Patients who achieved CR+good PR(Deauville score 4) after the rescue therapy will be consolidated with ASCT,and those remain in PR(Deauville score 5) will receive other rescue treatments(including ASCT+CAR T).

DETAILED DESCRIPTION:
Survival for patients with high risk aggressive B-cell lymphoma is still unsatisfied. Dose-intensified immunochemotherapy might improve the outcome. But for patients who could not achieve CR after the dose-intensified induction therapy, the prognosis is poor. The DLCL002 protocol is a total therapy which including induction therapy, rescue therapy and autologous stem cell transplantation. Patients eligible for the study will receive R-DA-EDOCH as the induction therapy and be evaluated by PET CT after the fourth cycle. Patients achieve CR at interim-PET(Deauville score 1-3) will receive either ASCT or the remaining 4 cycles of R-DA-EDOCH, while those achieve PR(Deauville score 4-5) will be rescued by two courses of R(2)-DHAP and then be revaluated by the second interim-PET. Patients who achieved CR+good PR(Deauville score 4) after the rescue therapy will be consolidated with ASCT,and those remain in PR(Deauville score 5) will receive other rescue treatments(including ASCT+CAR T).

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmed aggressive B-cell lymphoma with one of the following subtypes:

  1. diffuse large B-cell lymphoma, NOS with at least one poor prognostic factor as follows:

     1. aaIPI 2~3(≤60 years) or IPI 3~5(>60 years);
     2. double protein expression lymphoma(IHC MYC≥40% and BCL2≥50%） with Ann Arbor stage of III~IV or aaIPI 2~3 or IPI 3~5;
     3. CD5+ DLBCL.
  2. high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements;
  3. high-grade B-cell lymphoma, NOS
  4. transformed lymphoma(no prior treatment)
* Age 18 to 65 years
* ECOG-PS: 0~2
* Life-expectancy > 3 months

Exclusion Criteria:

* Patients with central nerves system involvement
* HIV positivity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2019-01-21 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
PFS | From the date of the start of treatment until the date of first documented progression, relapse or death from any cause, whichever came first, assessed up to 2 years.
  progression free survival

SECONDARY OUTCOMES:
ORR | up to 3 months after the end of the therapy
  objective response rate
EFS | From the date of the start of treatment until the date of the ﬁrst adverse event (i.e. disease progression, relapse, diagnosis of a secondary malignancy, institution of a new anticancer treatment, any cause of death), assessed up to 2 years.
  event free survival
OS | From the date of the start of treatment until the date of death from any cause, assessed up to 2 years.
  overall survival
CRR | up to 3 months after the end of the therapy
  complete response rate

CONTACTS AND LOCATIONS:
Overall Officials: Dehui Zou, Dr., Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (6):
- China (6):
  - Hunan Cancer Hospital, Changsha, Hunan
  - the First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - the First Affiliated Hospital of Jilin University, Changchun, Jilin
  - the Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Qingdao Central Hospital, Qingdao, Shandong
  - Institute of Hematology & Blood Diseases Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: Undecided